CLINICAL TRIAL: NCT00673296
Title: Intravitreal Injection of Bevacizumab and Gas for Diabetic Premacular Hemorrhage With Active Fibrovascular Proliferation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chung-May Yang, M.D., Natinal Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200711050R
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-04

CONDITIONS: Diabetic Retinopathy With Premacular Hemorrhage
Keywords: Bevacizumab; Diabetic premacular hemorrhage; Intravitreal gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Other): Patients receive intravitreal injection of bevacizumab (1.25 mg in 0.05 mL) and C3F8 (0.2-0.3 mL)
  Interventions: Drug: Intravitreal Bevacizumab

INTERVENTIONS:
Drug: Intravitreal Bevacizumab — Intravitreal injection of bevacizumab (1.25 mg in 0.05 mL) and C3F8 (0.2-0.3 mL)

SUMMARY:
Diabetic premacular hemorrhage occurs when blood from preretinal neovascular tissue is entrapped between the retina and the posterior hyaloid in the macular area. It may occur spontaneously or secondary to traction from a localized posterior vitreous detachment. This complication may greatly disturb the central vision and may be an important stimulant of fibrovascular proliferation.

Bevacizumab (Avastin, Genentech, Inc.) is a humanized monoclonal antibody against vascular endothelial growth factor (VEGF), which has been used to treat a variety of neovascular ocular diseases. In proliferative diabetic retinopathy, intravitreal bevacizumab has been shown to induce prompt regression of neovascularization and may enhance resolution of vitreous hemorrhage.

In this study, we propose that simultaneous intravitreal injection of gas and bevacizumab may be a useful treatment option in diabetic premacular hemorrhage with active fibrovascular tissue. In this procedure, gas is used to displace the blood while bevacizumab may render the neovascularization less active to decrease the likelihood of recurrent hemorrhage.

DETAILED DESCRIPTION:
In this study, consecutive cases of acute diabetic premacular hemorrhage and active fibrovascular proliferation will receive intravitreal injection of bevacizumab (1.25 mg in 0.05 mL) and C3F8 (0.2-0.3 mL) during the same setting. Before intravitreal injection, all patients should either have complete panretinal photocoagulation (PRP) treatment or PRP to the peripheral retina. After treatment, patients will maintain a prone position for three days and be followed at regular interval. After vitreous clear-up, further supplementary PRP extending beyond equator will be done. Snellen best-corrected visual acuity measurements, intraocular pressure, slit-lamp examination and non-contact lens biomicroscopic examination will be performed before treatment and at each follow-up visit. Data including the extent of premacular hemorrhage, and the interval between the treatment and clearing of premacular hemorrhage will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Acute diabetic premacular hemorrhage and minor active fibrovascular proliferation

Exclusion Criteria:

* Anticoagulant therapy
* Blood diseases associated with abnormal coagulation
* Proliferative retinopathy severe enough to warrant vitrectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Interval between the treatment and clearing of premacular hemorrhage | Before treatment, weekly after the treatment, and monthly after hemorrhage reabsorption

SECONDARY OUTCOMES:
Snellen best-corrected visual acuity measurements, intraocular pressure, slit-lamp examination and non-contact lens biomicroscopic examination. | Before treatment, weekly after the treatment, and monthly after hemorrhage reabsorption

CONTACTS AND LOCATIONS:
Overall Officials: Chung May Yang, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Michels RG. Proliferative diabetic retinopathy: pathophysiology of extraretinal complications and principles of vitreous surgery. Retina. 1981;1(1):1-17. PMID 15633404
- [Background] Yang CM, Chen MS. Tissue plasminogen activator and gas for diabetic premacular hemorrhage. Am J Ophthalmol. 2000 Mar;129(3):393-4. doi: 10.1016/s0002-9394(99)00393-1. PMID 10704565
- [Background] Chung J, Kim MH, Chung SM, Chang KY. The effect of tissue plasminogen activator on premacular hemorrhage. Ophthalmic Surg Lasers. 2001 Jan-Feb;32(1):7-12. PMID 11195747
- [Background] Lynch SS, Cheng CM. Bevacizumab for neovascular ocular diseases. Ann Pharmacother. 2007 Apr;41(4):614-25. doi: 10.1345/aph.1H316. Epub 2007 Mar 13. PMID 17355998
- [Background] Spaide RF, Fisher YL. Intravitreal bevacizumab (Avastin) treatment of proliferative diabetic retinopathy complicated by vitreous hemorrhage. Retina. 2006 Mar;26(3):275-8. doi: 10.1097/00006982-200603000-00004. PMID 16508426
- [Background] Verheul HM, Jorna AS, Hoekman K, Broxterman HJ, Gebbink MF, Pinedo HM. Vascular endothelial growth factor-stimulated endothelial cells promote adhesion and activation of platelets. Blood. 2000 Dec 15;96(13):4216-21. PMID 11110694
- [Background] Arevalo JF, Maia M, Flynn HW Jr, Saravia M, Avery RL, Wu L, Eid Farah M, Pieramici DJ, Berrocal MH, Sanchez JG. Tractional retinal detachment following intravitreal bevacizumab (Avastin) in patients with severe proliferative diabetic retinopathy. Br J Ophthalmol. 2008 Feb;92(2):213-6. doi: 10.1136/bjo.2007.127142. Epub 2007 Oct 26. PMID 17965108
- [Derived] Shih CW, Yang CM, Chen MS, Wang TJ. Intravitreal injection of bevacizumab and gas for diabetic premacular hemorrhage with active fibrovascular proliferation. Graefes Arch Clin Exp Ophthalmol. 2008 Nov;246(11):1547-51. doi: 10.1007/s00417-008-0902-8. Epub 2008 Aug 6. PMID 18682973